Official title:comparative study of nonintubated uniport thoracoscopic surgery using thoracic paravertebral nerve block versus intercostal nerve block for peripheral solitary pulmonary nodule patients

NCT number:03086213

Document date: April 7,2020

Statistical analysis plan

Updated:April 7,2020

The evaluation of the pain scale of the enrolled subjects was performed using the visual analog score (VAS) and graded between 0 (no pain) and 10 (severe pain) after the operation. The study phase lasted 48 hours, and the data collection was performed by a person not involved in the study (ward nurse assigned beforehand) and the VAS was entered in a case report form. The following parameters were assessed: (1) quantity of intravenous drugs administered such as propofol, remifentanil, and dexmedetomidine; (2) adverse events related to puncture, including bleeding; hematoma; nerve injury; postoperative pain scores at 1, 6, 24, and 48 hours; requirement for rescue analgesia (morphine); adverse effects of the analgesia procedure, including respiratory depression, pneumothorax, cardiotoxicity, sedation, urinary retention, nausea, vomiting, and pruritus. Descriptive statistics are shown as means ± SD for continuous data and as number and percentage for categorical data. The two-sample t-test was employed for statistical analysis of continuous variables and Fisher exact test was used for the statistical analysis of categorical variables such as sex. All data analyses were performed using SPSS 22.0 (Chicago, IL) and all statistical tests were two-sided. Statistical significance was defined as a p value of less than 0.05